CLINICAL TRIAL: NCT02307097
Title: Randomised Controlled Trial of Cognitive-Behavioural Bibliotherapy (CBB) for Social Anxiety Disorder as a Prelude to High-Intensity Cognitive-Behavioural Therapy (CBT) in a Local IAPT Service.
Brief Title: RCT of Bibliotherapy for Social Anxiety Disorder as a Prelude to CBT in IAPT
Acronym: RCT of CBB/CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solent NHS Trust (Other Government)
Collaborators: University of Oxford (Other); Talking Change (Solent NHS Trust) (Unknown); Constable & Robinson (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-OxCADAT-2014
Record Dates: First submitted 2014-11-30; First posted 2014-12-04 (Estimated); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Bibliotherapy; Social Anxiety Disorder; Cognitive Behavioral Therapy
Keywords: Randomised Controlled Trial; Cognitive-Behavioural Bibliotherapy; Social Anxiety Disorder; Cognitive-Behavioural Therapy; IAPT
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CBB (Experimental)
  Interventions: Procedure: Cognitive-Behavioural Bibliotherapy
- CBT (Experimental)
  Interventions: Procedure: Cognitive-Behavioural Therapy
- WAIT (Active Comparator)
  Interventions: Other: WAIT

INTERVENTIONS:
Procedure: Cognitive-Behavioural Bibliotherapy
  Arms: CBB
Procedure: Cognitive-Behavioural Therapy
  Arms: CBT
Other: WAIT
  Arms: WAIT

SUMMARY:
The efficacy of high-intensity Cognitive-Behavioural Therapy (CBT) for social anxiety disorder is well established (Mayo-Wilson et al., 2014) and it is recommended by the National Institute of Health and Clinical Excellence (NICE) as the first-line psychological intervention for social anxiety disorder. The treatment aims to modify several maintenance factors (e.g., self-focused attention) that are specified in cognitive models of social anxiety disorder (e.g., Clark & Wells, 1995).

Cognitive-behavioural self-help treatments for social anxiety disorder have been developed to overcome various accessibility issues (e.g., long wait-lists, and the patient's need to avoid social situations, etc) associated with high-intensity CBT (Abramowitz et al., 2009; Carlbring et al., 2007) but a recent network meta-analysis (Mayo-Wilson et al., 2014) identified the former as less cost-effective than the later and thus, they are not recommended as standalone treatments.

However, the potential benefit of cognitive-behavioural self-help treatments for social anxiety disorder within a stepped-care recovery model as a prelude to high-intensity CBT has not been formally evaluated.

The aim of this study is to evaluate a seminal Cognitive-Behavioural Bibliotherapy* (CBB; "pure self-help" book) - 'Overcoming Social Anxiety & Shyness' (Butler, 2009) - for patients with social anxiety disorder while on the wait-list for high-intensity CBT within an Improving Access to Psychological Therapies (IAPT) service, and to determine if some patients recover from CBB alone or whether there may be a reduction in the average number of high-intensity CBT sessions for those patients who subsequently require further treatment.

The study is funded by Constable & Robinson, Kellogg College (University of Oxford) and Talking Change (Solent NHS Trust).

* The Reading Well Books on Prescription scheme with funding from the Arts Council England enables general practitioners (GPs) and mental health professionals to prescribe seminal CBBs for patients with mood and anxiety disorders. The books are accessed free of charge via local libraries. The scheme works within NICE guidelines and it is support by the Royal Colleges of GPs, Nursing and Psychiatrists, the British Association for Behavioural and Cognitive Psychotherapies and the Department of Health through its IAPT programme.

DETAILED DESCRIPTION:
P A R T I C I P A N T S

Patients will be recruited within an Improving Access to Psychological Therapies (IAPT) service: 'Talking Change' (Portsmouth). Advertisement for the study will be distributed locally, through social media and via the 'Talking Change' Internet website.

It is generally accepted that social anxiety disorder is a chronic condition and significant change in the wait-list does not occur. Hence, because the study aims to explore predicators of treatment response, a priori power analyses determined that approximately 114 patients randomly assigned for twelve-weeks at a ratio of 2:1 would provide sufficient power for statistical analyses; seventy-six and thirty-eight patients in the Cognitive-Behavioural Bibliotherapy (CBB) and wait-list control (WAIT) group, respectively.

Randomisation will be conducted by someone unassociated with the study using sealed envelopes.

M E A S U R E S

Risk Assessment:

An IAPT-standard risk assessment will be utilised.

Diagnostic measures:

Diagnostic interviews will use a combination of the Anxiety and Related Disorders Interview Schedule (ADIS-5; Brown & Barlow, 2014) for the Diagnostic and Statistical Manual of Mental Disorders (5th ed.; DSM-5; American Psychiatric Association, 2013) to identify social anxiety disorder and the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders (4th ed.; DSM-4; American Psychiatric Association, 1994) Axis I disorders (SCID-I; First, Spitzer, Gibbon and Williams, 1995) and Axis II disorders (SCID-II; First, Gibbon, Spitzer, Williams and Benjamin, 1997). All patients will be assessed with the social anxiety disorder module of the ADIS, the overview and screener modules of the SCID-I, and the screener questionnaire for SCID-II. If the SCID-I screener module indicates that another Axis I disorder might be present, the SCID-I module for that disorder will also be administered. The same applies to the screener questionnaire for the SCID-II. However, regardless of screening responses, all patients will also be assessed with the avoidant personality disorder section of the SCID-II.

The Social Phobia Inventory (SPIN; Connor, 2000) will assess the main spectrum of social anxiety disorder such as fear, avoidance, and physiological symptoms.

The Adult Reading Test (ART; Everatt, Brooks, & Fidler, 2004) will assess reading accuracy, reading comprehension, speed of reading and speed of writing.

Primary measures (CBB, CBT and WAIT groups):

IAPT Standard Minimum Data Set (MDS): The brief versions of the Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001) and the Generalised Anxiety Disorder Questionnaire (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006) will assess mood and generalised anxiety, respectively. The Work and Social Adjustment Scale (WSAS; Marks, 1986) will assess functional impairment attributable to an identified problem. The Phobia Scales is a non-validated phobia screener of social phobia, panic disorder/agoraphobia, and specific phobia avoidance.

The Social Phobia Inventory (SPIN; Connor, 2000) will assess the main spectrum of social anxiety disorder such as fear, avoidance, and physiological symptoms.

The Social Participation & Satisfaction Questionnaire (SPSQ; Alden & Taylor, 2011) will assess the degree by which the participant is participating is social activity, and relationship satisfaction.

Secondary measures (CBB, CBT and WAIT groups):

The self-report version of the Liebowitz Social Anxiety Scale (LSAS-SR; Baker, Heinrich, Kim, & Hofmann, 2002; Liebowitz, 1987) will assess social anxiety and the frequency of avoidance.

The Self-Focused Attention Scale (SFA; Bögels, Alberts, & de Jong, 1996) will assess the degree by which the participant engages in self-focused attention.

The Social Behaviour Questionnaire (SBQ; Clark et al., 2006) will assess the frequency by which the participant engages in a range of common safety-seeking behaviours.

The Social Phobia Cognitions Questionnaire (SPC; Clark et al., 2006) will assess the frequency and belief ratings for a range of typical cognitions in social anxiety.

The Anticipatory Processing Questionnaire (APQ; Vassilopoulos, 2004) and the Post-Event Processing Questionnaire-Revised (PEPQ-R; McEvoy & Kingsep, 2006) will assess the degree by which the participant engages in pre- and post-event rumination.

Weekly measures [CBB and CBT groups only]:

IAPT Standard Minimum Data Set (MDS): The brief versions of the Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001) and the Generalised Anxiety Disorder Questionnaire (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006) will assess mood and generalised anxiety, respectively. The Work and Social Adjustment Scale (WSAS; Marks, 1986) is a self-report scale of functional impairment attributable to an identified problem. The Phobia Scales is a non-validated phobia screener of social phobia, panic disorder/agoraphobia, and specific phobia avoidance.

The self-report version of the Liebowitz Social Anxiety Scale (LSAS-SR; Baker, Heinrich, Kim, & Hofmann, 2002; Liebowitz, 1987) will be administrated weekly to assess social anxiety and the frequency of avoidance.

The Social Phobia Inventory (SPIN; Connor, 2000) will assess the main spectrum of social anxiety disorder such as fear, avoidance, and physiological symptoms.

A written answer to the question "What have I learnt?" will assess treatment compliance.

Qualitative measure (if received CBB):

A semi-structured interview of patients' experiences.

Other measures:

The number of high-intensity CBT sessions required following CBB will be recorded.

P R O C E D U R E

Patients will engage with a brief telephone Triage Assessment of their presenting problems and will complete the primary measures to assess symptoms of social anxiety, depression, generalised anxiety, phobia avoidance, general functioning, and social functioning.

Patients will be "stepped-up" to a full face-to-face Step Three Assessment of their presenting problems if their condition is chronic and cannot be appropriately treated with a Step 2 intervention. Thus, potential cases of social anxiety disorder who score within the clinical range (≥19 points) on the SPIN (Connor, 2000) will be "stepped-up". All other cases will be offered alternative treatment within the service or referred elsewhere as required.

Patients will complete the diagnostic measures to determine social anxiety disorder, a measure of reading and writing ability, the primary measures again, and the secondary measures to assess the maintenance factors that are specified in cognitive models of social anxiety disorder (e.g., Clark & Wells, 1995). Patients who do not meet the inclusion criteria will be offered alternative treatment within the service or referred elsewhere as required.

Patients who consent to their participation in the study will be randomly allocated to CBB or WAIT for twelve weeks. The wait-list group will begin high-intensity CBT at postWAIT.

Patients who are not "CBB responders"* will receive high-intensity CBT at postCBB whereas those who are will be discharged from the service, offered alternative treatment within the service if "caseness"** remains, or referred elsewhere as required.

The primary and secondary measures will be completed again at preCBB-WAIT-CBT, midCBB-WAIT-CBT, postCBB-WAIT-CBT, and CBB-CBT one-month follow-up. The CBB and CBT group will complete the primary measures weekly complete and weekly measures of social anxiety. The CBB group only will complete a weekly measure of treatment compliance.

Patients will the complete diagnostic measures to determine social anxiety disorder, the primary measures and the secondary measures again at postCBB-WAIT-CBT and CBB-CBT one-month follow-up. A qualitative measure of patients' experiences of treatment will be obtained at postCBB, and postCBT if they previously received CBB.

Patients will be notified when measures must be completed; most of which are completed online a secure and encrypted Internet website and some of which are completed face-to-face.

The CBB group will be provided with a self-help book ('Overcoming Social Anxiety & Shyness'; Butler, 2009) by local libraries and encouraged to work through in a twelve-week period. A suggested timetable for completing the "pure self-help" treatment will be provided. Clinical or non-clinical contact will not be provided. The CBT group will receive up to fourteen face-to-face sessions of high-intensity CBT at their local clinic.

Patients will be provided the Chief Investigator's contact details should they wish to discuss any aspect of the study or if they become distressed. If patients' risk status should change during the trail they will be instructed to contact the Chief Investigator immediately.

At the end of study all patients will be discharged from the service, offered alternative treatment within the service if "caseness" remains, or referred elsewhere as required.

* Those patients who have a statistically reliable improvement that place their mean LSAS-SR score within the range (mean ± two standard deviations) of the non-clinical population mean, who score ≤ 18 points on the SPIN (Connor, 2000), and who no longer meet full DSM-V criteria for social anxiety disorder (APA, 2013) will be "CBB responders" (i.e., a clinically significant change; see Jacobson & Truax, 1991). The non-clinical population mean will be based on Fresco et al.'s (2001) non-anxious control group.

** The IAPT programme defines "caseness" as ≤ 9 points on the PHQ-9 (Kroenke, Spitzer, & Williams, 2001) and ≤ 7 points on the GAD-7 (Spitzer, Kroenke, Williams, & Löwe, 2006).

ELIGIBILITY:
Inclusion criteria:

* ≥ 18 years of age;
* ≥ 19 points on the Social Phobia Inventory (SPIN; Connor, 2000);
* Meets full Diagnostic and Statistical Manual of Mental Disorders (5th ed.;
* DSM-5; American Psychiatric Association, 2013) criteria for social anxiety disorder;
* Social anxiety is the primary disorder requiring treatment;
* Sufficient reading and writing ability (cut-off to be decided);
* English is first language;
* Stable dose of antidepressant medication for at least two months.

Patients who do not meet the inclusion criteria will be offered alternative treatment within the service or referred elsewhere as required.

Exclusion criteria:

* If co-morbidity present, social anxiety disorder is not the primary problem;
* Another disorder (e.g., depression) requires urgent treatment in it's own right;
* Past or present history of psychosis, borderline personality disorder, or bipolar disorder;
* Risk to themselves or others; Drug and alcohol misuse;
* Previous high-intensity Cognitive-Behavioural Therapy (CBT) for social anxiety disorder;
* On-going psychological therapy;
* Engaging in another research trial;
* Psychotropic medication.

Patients who meet the exclusion criteria will be offered alternative treatment within the service or referred elsewhere as required.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
IAPT Standard Minimum Data Set (MDS) | 2 minutes
  The brief versions of the Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001) and the Generalised Anxiety Disorder Questionnaire (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006) will assess mood and generalised anxiety, respectively. The Work and Social Adjustment Scale (WSAS; Marks, 1986) will assess functional impairment attributable to an identified problem. The Phobia Scales is a non-validated phobia screener of social phobia, panic disorder/agoraphobia, and specific phobia avoidance.
The Social Phobia Inventory (SPIN; Connor, 2000) | 2 minutes
  The SPIN will assess the main spectrum of social anxiety disorder such as fear, avoidance, and physiological symptoms.
The Social Participation & Satisfaction Questionnaire (SPSQ; Alden & Taylor, 2011) | 2 minutes
  The SPSQ will assess the degree by which the participant is participating is social activity, and relationship satisfaction.

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS-SR; Baker, Heinrich, Kim, & Hofmann, 2002; Liebowitz, 1987) | 2 minutes
  The self-report version of the LSAS-SR will assess social anxiety and the frequency of avoidance.
Self-Focused Attention Scale (SFA; Bögels, Alberts, & de Jong, 1996) | 2 minutes
  The SFA will assess the degree by which the participant engages in self-focused attention.
Social Behaviour Questionnaire (SBQ; Clark et al., 2006) | 2 minutes
  The SBQ will assess the frequency by which the participant engages in a range of common safety-seeking behaviours.
Social Phobia Cognitions Questionnaire (SPC; Clark et al., 2006) | 2 minutes
  The SPC will assess the frequency and belief ratings for a range of typical cognitions in social anxiety.
Anticipatory Processing Questionnaire (APQ; Vassilopoulos, 2004) and Post-Event Processing Questionnaire-Revised (PEPQ-R; McEvoy & Kingsep, 2006) | 2 minutes
  The APQ and PEPQ-R will assess the degree by which the participant engages in pre- and post-event rumination.

OTHER OUTCOMES:
A written answer to the question "What have I learnt?" will assess treatment compliance. | 5 minutes
A semi-structured interview of patients' experiences. | 10 minutes
The number of high-intensity CBT sessions required following CBB will be recorded. | 0 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Miles D Wrightman, MSc, Principal Investigator — University of Oxford; Professor David M Clark, DPhil, Study Director — University of Oxford
Locations (1):
- Talking Change (Solent NHS Trust), Portsmouth, Hampshire, United Kingdom

REFERENCES:
- [Background] Abramowitz JS, Moore EL, Braddock AE, Harrington DL. Self-help cognitive-behavioral therapy with minimal therapist contact for social phobia: a controlled trial. J Behav Ther Exp Psychiatry. 2009 Mar;40(1):98-105. doi: 10.1016/j.jbtep.2008.04.004. Epub 2008 Apr 26. PMID 18514614
- [Background] Clark, D. M., & Wells, A. (1995). A cognitive model of social phobia. In R. Heimberg, M. Liebowitz, D. A. Hope, & F. R. Schneier (Eds.), Social phobia: Diagnosis, assessment, and treatment (pp. 69-93). New York: Guilford Press.
- [Background] Butler, G. (2009). Overcoming Social Anxiety & Shyness. London: Robinson Publishing.
- [Background] Carlbring P, Gunnarsdottir M, Hedensjo L, Andersson G, Ekselius L, Furmark T. Treatment of social phobia: randomised trial of internet-delivered cognitive-behavioural therapy with telephone support. Br J Psychiatry. 2007 Feb;190:123-8. doi: 10.1192/bjp.bp.105.020107. PMID 17267928
- [Background] Mayo-Wilson E, Dias S, Mavranezouli I, Kew K, Clark DM, Ades AE, Pilling S. Psychological and pharmacological interventions for social anxiety disorder in adults: a systematic review and network meta-analysis. Lancet Psychiatry. 2014 Oct;1(5):368-76. doi: 10.1016/S2215-0366(14)70329-3. Epub 2014 Oct 7. PMID 26361000
- See also: The Oxford Centre for Anxiety Disorders and Trauma (University of Oxford) — http://oxcadat.psy.ox.ac.uk
- See also: Constable & Robinson — http://www.constablerobinson.com